CLINICAL TRIAL: NCT01740362
Title: Phase 1, Open-Label Study To Evaluate Single Dose Pharmacokinetics, Safety And Tolerability Of CP-690,550 In Patients With Impaired Renal Function
Brief Title: Pharmacokinetics Of CP-690,550 In Patients With Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: A3921006
Record Dates: First submitted 2012-10-16; First posted 2012-12-04 (Estimated); Results first posted 2013-01-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2012-12

CONDITIONS: Renal Impairment
Keywords: CP-690; 550; pharmacokinetics; renal impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy volunteers (Other): Healthy volunteers
  Interventions: Drug: CP-690,550
- Mild renal impairment (Experimental): patients with mild (>50 and ≤80 mL/min) renal impairment
  Interventions: Drug: CP-690,550
- Moderate renal impairment (Experimental): patients with moderate (≥30 and ≤50 mL/min) renal impairment
  Interventions: Drug: CP-690,550
- severe renal impairment (Experimental): patients with severe (<30 mL/min) renal impairment
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: CP-690,550 — 10 mg (2 x 5 mg tablets), single dose
  Arms: Healthy volunteers
Drug: CP-690,550 — 10 mg (2 x 5 mg tablets), single dose
  Arms: Mild renal impairment
Drug: CP-690,550 — 10 mg (2 x 5 mg tablets), single dose
  Arms: Moderate renal impairment
Drug: CP-690,550 — 10 mg (2 x 5 mg tablets), single dose
  Arms: severe renal impairment

SUMMARY:
A study to evaluate the pharmacokinetics of CP-690,550 in subjects with mild, moderate or severe renal impairment, who do not require hemodialysis, compared to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with normal renal function: Subjects must be healthy with estimated creatinine clearance >80 mL/min
* Subjects with renal impairment: Subjects should be in good general health commensurate with the population with chronic kidney disease

Exclusion Criteria:

* Kidney transplant patients
* Subjects with any condition possibly affecting drug absorption
* Subjects with malignancies with the exception of adequately treated basal cell carcinoma of the skin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-10; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Minneapolis, Minnesota

REFERENCES:
- [Derived] Krishnaswami S, Chow V, Boy M, Wang C, Chan G. Pharmacokinetics of tofacitinib, a janus kinase inhibitor, in patients with impaired renal function and end-stage renal disease. J Clin Pharmacol. 2014 Jan;54(1):46-52. doi: 10.1002/jcph.178. Epub 2013 Sep 30. PMID 24030917
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921006&StudyName=Pharmacokinetics%20Of%20CP-690%2C550%20In%20Patients%20With%20Impaired%20Renal%20Function%20

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 (Normal Renal Function): Participants with normal renal function who had creatinine clearance greater than (>) 80 milliliter/minute (mL/min), received single oral dose of CP-690,550 tablet 10 milligram (mg) orally.
- CP-690,550 (Mild Renal Insufficiency): Participants with mild renal insufficiency who had creatinine clearance >50 mL/min but less than or equal to (=<) 80 mL/min, received single oral dose of CP-690,550 tablet 10 mg orally.
- CP-690,550 (Moderate Renal Insufficiency): Participants with moderate renal insufficiency who had creatinine clearance >=30 mL/min but =<50 mL/min, received single oral dose of CP-690,550 tablet 10 mg orally.
- CP-690,550 (Severe Renal Insufficiency): Participants with severe renal insufficiency who had creatinine clearance <30 mL/min, received single oral dose of CP-690,550 tablet 10 mg orally.
Period: Overall Study
Arm/Group | CP-690,550 (Normal Renal Function) | CP-690,550 (Mild Renal Insufficiency) | CP-690,550 (Moderate Renal Insufficiency) | CP-690,550 (Severe Renal Insufficiency)
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CP-690,550 (Normal Renal Function) | CP-690,550 (Mild Renal Insufficiency) | CP-690,550 (Moderate Renal Insufficiency) | CP-690,550 (Severe Renal Insufficiency) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 50.8 (9.7) | 61.2 (2.8) | 53.5 (11.1) | 59.0 (14.6) | 56.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4 | 3 | 11
  Male | 4 | 4 | 2 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)]
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: 0 (Pre-dose), 0.5, 1, 1.5, 2, 4, 8, 10, 12, 16, 24, 48 hours post-dose
Population: Analysis set included all participants who received study medication.
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | CP-690,550 (Normal Renal Function) | CP-690,550 (Mild Renal Insufficiency) | CP-690,550 (Moderate Renal Insufficiency) | CP-690,550 (Severe Renal Insufficiency)
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram*hour/milliliter (ng*hr/mL) | 268 (71.5) | 370 (109) | 396 (154) | 615 (214)
Statistical Analysis 1: Comparison: CP-690,550 (Normal Renal Function) vs CP-690,550 (Mild Renal Insufficiency); 1 way Analysis of Variance (ANOVA) on natural log-transformed AUC(0-∞) analyzed using linear model with degrees of renal impairment(creatinine clearance[CLcr, discrete]) evaluated using blood samples collected at screening as fixed effect. Statistical Analysis System (SAS) mixed procedure (PROC MIXED) was used. Anti-log of adjusted mean difference (CP-690,550[mild renal insufficiency] - CP-690,550[normal renal function]), 90% confidence interval (CI) were taken to estimate mean ratio and 90% CI; Test type: Superiority or Other; Ratio of adjusted geometric means = 137.26, 90% CI 2-sided [96.77 to 194.69]
Statistical Analysis 2: Comparison: CP-690,550 (Normal Renal Function) vs CP-690,550 (Moderate Renal Insufficiency); One way ANOVA on natural log-transformed AUC (0 - ∞) were analyzed using linear model containing degrees of renal impairment (CLcr, discrete) calculated using blood samples collected at screening as fixed effects. SAS procedure PROC MIXED was used for analysis. Anti-log of the adjusted mean difference (CP-690,550 [moderate renal insufficiency] - CP-690,550 [normal renal function]) and its corresponding 90% CI were taken to estimate the mean ratio and corresponding 90% CI; Test type: Superiority or Other; Ratio of adjusted geometric means = 142.59, 90% CI 2-sided [100.53 to 202.24]
Statistical Analysis 3: Comparison: CP-690,550 (Normal Renal Function) vs CP-690,550 (Severe Renal Insufficiency); One way ANOVA on natural log-transformed AUC (0 - ∞) were analyzed using linear model containing degrees of renal impairment (CLcr, discrete) calculated using blood samples collected at screening as fixed effects. SAS procedure PROC MIXED was used for analysis. Anti-log of the adjusted mean difference (CP-690,550 [severe renal insufficiency] - CP-690,550 [normal renal function]) and its corresponding 90% CI were taken to estimate the mean ratio and corresponding 90% CI; Test type: Superiority or Other; Ratio of adjusted geometric means = 222.71, 90% CI 2-sided [157.02 to 315.89]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0 (Pre-dose), 0.5, 1, 1.5, 2, 4, 8, 10, 12, 16, 24, 48 hours post-dose
Population: Analysis set included all participants who received study medication.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 (Normal Renal Function) | CP-690,550 (Mild Renal Insufficiency) | CP-690,550 (Moderate Renal Insufficiency) | CP-690,550 (Severe Renal Insufficiency)
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL | 94.2 (25.3) | 87.3 (23.2) | 104 (47.5) | 111 (28.6)
Statistical Analysis 1: Comparison: CP-690,550 (Normal Renal Function) vs CP-690,550 (Mild Renal Insufficiency); One way ANOVA on natural log-transformed Cmax were analyzed using linear model containing degrees of renal impairment (CLcr, discrete) calculated using blood samples collected at screening as fixed effects. SAS procedure PROC MIXED was used for analysis. Anti-log of the adjusted mean difference (CP-690,550 [mild renal insufficiency] - CP-690,550 [normal renal function]) and its corresponding 90% CI were taken to estimate the mean ratio and corresponding 90% CI; Test type: Superiority or Other; Ratio of adjusted geometric mean = 93.15, 90% CI 2-sided [67.22 to 129.06]
Statistical Analysis 2: Comparison: CP-690,550 (Normal Renal Function) vs CP-690,550 (Moderate Renal Insufficiency); One way ANOVA on natural log-transformed Cmax were analyzed using linear model containing degrees of renal impairment (CLcr, discrete) calculated using blood samples collected at screening as fixed effects. SAS procedure PROC MIXED was used for analysis. Anti-log of the adjusted mean difference (CP-690,550 [moderate renal insufficiency] - CP-690,550 [normal renal function]) and its corresponding 90% CI were taken to estimate the mean ratio and corresponding 90% CI; Test type: Superiority or Other; Ratio of adjusted geometric mean = 104.17, 90% CI 2-sided [75.18 to 144.34]
Statistical Analysis 3: Comparison: CP-690,550 (Normal Renal Function) vs CP-690,550 (Severe Renal Insufficiency); One way ANOVA on natural log-transformed Cmax were analyzed using linear model containing degrees of renal impairment (CLcr, discrete) calculated using blood samples collected at screening as fixed effects. SAS procedure PROC MIXED was used for analysis. Anti-log of the adjusted mean difference (CP-690,550 [severe renal insufficiency] - CP-690,550 [normal renal function]) and its corresponding 90% CI were taken to estimate the mean ratio and corresponding 90% CI; Test type: Superiority or Other; Ratio of adjusted geometric mean = 117.65, 95% CI 2-sided [84.91 to 163.02]

3. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0 (Pre-dose), 0.5, 1, 1.5, 2, 4, 8, 10, 12, 16, 24, 48 hours post-dose
Population: Analysis set included all participants who received study medication.
Measure: Median (Full Range); unit: hours
Arm/Group | CP-690,550 (Normal Renal Function) | CP-690,550 (Mild Renal Insufficiency) | CP-690,550 (Moderate Renal Insufficiency) | CP-690,550 (Severe Renal Insufficiency)
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours | 0.75 [0.50 to 1.50] | 1.00 [0.50 to 1.50] | 0.75 [0.50 to 2.00] | 0.75 [0.50 to 1.50]

4. Primary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (Pre-dose), 0.5, 1, 1.5, 2, 4, 8, 10, 12, 16, 24, 48 hours post-dose
Population: Analysis set included all participants who received study medication.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CP-690,550 (Normal Renal Function) | CP-690,550 (Mild Renal Insufficiency) | CP-690,550 (Moderate Renal Insufficiency) | CP-690,550 (Severe Renal Insufficiency)
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours | 2.37 (0.363) | 2.83 (0.857) | 2.88 (0.653) | 3.77 (0.480)

5. Primary Outcome: Renal Clearance (CL R)
Description: Renal clearance is the volume of plasma from which the drug is completely removed by the kidney in a given amount of time.
Time Frame: 0 (Pre-dose) to 12 hours post-dose, 12 to 24 hours post-dose
Population: Analysis set included all participants who received study medication.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | CP-690,550 (Normal Renal Function) | CP-690,550 (Mild Renal Insufficiency) | CP-690,550 (Moderate Renal Insufficiency) | CP-690,550 (Severe Renal Insufficiency)
Number analyzed (Participants) | 6 | 6 | 6 | 6
mL/min | 113 (16.2) | 84.7 (28.7) | 27.4 (15.9) | 19.9 (7.52)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-690,550 (Normal Renal Function) | CP-690,550 (Mild Renal Insufficiency) | CP-690,550 (Moderate Renal Insufficiency) | CP-690,550 (Severe Renal Insufficiency)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 3/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 (Normal Renal Function) (N=6) | CP-690,550 (Mild Renal Insufficiency) (N=6) | CP-690,550 (Moderate Renal Insufficiency) (N=6) | CP-690,550 (Severe Renal Insufficiency) (N=6)
Hypertension (Cardiac disorders) | 0 | 0 | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.